CLINICAL TRIAL: NCT00575107
Title: A System for Lengthening Contraction Training of Muscle
Acronym: LCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: BioLogic Engineering, Inc. (Industry)
Responsible Party: Neil Alexander, MD, Department of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-0319
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSC-VLC (Experimental): velocity-controlled variable resistance, lengthening contraction
  Interventions: Other: Exercise
- SC (Active Comparator): Constant weight shortening contraction
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Velocity-controlled variable resistance protocols enable trainees to load their muscles more optimally along the entire ROM in either or both of the shortening (VSC) and lengthening (VLC) phases of a training repetition
  Arms: VSC-VLC
Other: Exercise — Standard training of leg extension
  Arms: SC

SUMMARY:
Evaluation of a new exercise machine designed to improve strength and speed of movement in the leg muscles. Investigators are trying to learn whether a new training method results in greater strength improvements as compared to a traditional method.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* able to exercise 3 times per week for 16 weeks at Mobility Research Center

Exclusion Criteria:

* under- or overweight
* chronic disease that limits ability to exercise
* hips and legs limited by arthritis or pain
* presently engaged in a strenuous exercise program
* planned absence greater than one week.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Leg strength | 16 weeks

SECONDARY OUTCOMES:
Ability to rise from a chair | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Alexander, MD, Principal Investigator — University of Michigan
Locations (1):
- Mobility Research Center, Ann Arbor, Michigan, United States